CLINICAL TRIAL: NCT02436759
Title: A Randomized, Double-Masked, Placebo-Controlled Phase 3 Study of the Safety and Efficacy of RVL-1201 in the Treatment of Acquired Blepharoptosis
Brief Title: Study of the Safety and Efficacy of RVL-1201 in the Treatment of Acquired Blepharoptosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RVL Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVL-1201-201
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Acquired Blepharoptosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RVL-1201 (Experimental): RVL-1201 Ophthalmic Solution 0.1% 1 drop per eye QD for 6 weeks
  Interventions: Drug: RVL-1201
- RVL-1201 Vehicle Placebo (Placebo Comparator): RVL-1201 Ophthalmic Solution vehicle (placebo) 1 drop per eye QD for 6 weeks
  Interventions: Drug: RVL-1201 Vehicle Placebo

INTERVENTIONS:
Drug: RVL-1201 — RVL-1201 Ophthalmic Solution 0.1%
  Other Names: Oxymetazoline Hydrochloride Ophthalmic Solution 0.1%
  Arms: RVL-1201
Drug: RVL-1201 Vehicle Placebo — RVL-1201 Vehicle Placebo
  Other Names: RVL-1201 Ophthalmic Solution 0.1% Placebo
  Arms: RVL-1201 Vehicle Placebo

SUMMARY:
This is a Phase 3 study is to evaluate the safety and efficacy of RVL-1201 Ophthalmic Solution in the treatment of acquired blepharoptosis (ptosis) and to assess the safety and comfort of RVL-1201 Ophthalmic Solution for an extended dosing period of 6 weeks.

DETAILED DESCRIPTION:
Ptosis is experienced by approximately 12% of adults over the age of 50 . It is a unilateral or bilateral abnormal drooping of the upper eyelid that usually occurs from a partial or complete dysfunction of the muscle(s) that elevate the upper eyelid: the levator palpebrae superioris and/or Müller's muscle.

Treatment for acquired ptosis usually involves surgery, with risks of infection, bleeding, over or undercorrection, reduced vision, and lagophthalmos (inability to close the eyelids completely) or mechanical treatment e.g scleral contact lenses with a bar to lift the eyelid, eyelid ptosis crutches attached to glasses, or adhesive tape or putty to affix the upper eyelid to the supraorbital structures.

RVL-201 ophthalmic solution is being developed to provide a reversible pharmacologic option for patients with acquired ptosis who are not candidates for surgery or do not wish to undergo surgery.

The objective of this study is to evaluate the safety and efficacy of RVL-1201 ophthalmic solution in the treatment of acquired blepharoptosis and to assess the safety and comfort of RVL-1201 ophthalmic solution for an extended dosing period of 6 weeks. Subjects will be randomized (2:1) to one of 2 treatment arms and treated for 42 days:

* RVL-1201 0.1% one full drop in each eye QD in the morning (N = 100)
* RVL-1201 vehicle (placebo) 1 full drop per eye QD in the morning (N = 50)

Efficacy will be assessed with the LPFT, a validated visual field test using the HVF Analyzer and photographic measurement of MRD (the distance from the pupillary light reflex to the central margin of the upper lid) and PFD (the distance from the upper lid margin to the lower lid margin through the central visual axis). Safety assessment will include bilateral SLE/CFS, measurement of PD from external photographs, dilated ophthalmoscopy/fundus examination, tonometry, Snellen VA using recent correction, vital signs (BP/HR), and collection of adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age and older.
2. Presence of all of the following at Screening :

   a. Loss on a reliable LPFT of ≥ 8 points in the top 2 rows (LPFT Eligibility Score); subjects must see at least 9 total points in the top 4 rows (LPFT Total Score).

   i. This criteria must be met at both the Visit 1 Hour 0 (V1H0) and Visit 1 Hour 6 (V1H6) LPFT assessments

   ii. There must be ≤ 4 points of variance between the V1H0 and the V1H6 LPFT Eligibility Score;; AND

   b. The MRD, the distance from the central pupillary light reflex to the central margin of the upper lid, must be ≤ 2 mm (no visible central pupillary light reflex defaults to 0) in the same eye as Inclusion Criterion #2a

   AND

   c. Snellen visual acuity (VA) of 20/80 or better in the same eye as Inclusion Criteria #2a and #2b.
3. Presence of all of the following at Baseline:

   a. Loss on a reliable LPFT of ≥ 8 points in the top 2 rows (LPFT Eligibility Score) in the same eye as Inclusion Criterion #2a; subjects must see at least 9 total points in the top 4 rows (LPFT Total Score).

   i. This criteria must be met at the Visit 2 Hour 0 (V2H0) LPFT assessment. ii. There must be ≤ 4 points of variance between the V1H6 and the V2H0 LPFT Eligibility Score;

   AND

   b. Marginal Reflex Distance (MRD), the distance from the central pupillary light reflex to the central margin of the upper lid, must be ≤ 2 mm (no visible central pupillary light reflex defaults to 0) in the same eye as Inclusion Criterion #2a;

   AND

   c. Snellen VA of 20/80 or better in the same eye as Inclusion Criteria #2a and #2b.
4. Female subjects must be 1 year postmenopausal, surgically sterilized, or women of childbearing potential with a negative urine pregnancy test at Visit 1. Women of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.
5. Able to self-administer study medication or to have the study medication administered by a caregiver throughout the study period.
6. Subjects must be able to understand and sign an IRB approved informed consent form prior to participation in any study-related procedures.

Exclusion Criteria:

In either eye

1. Congenital ptosis.
2. Presence of either of the following:

   1. Pseudoptosis (upper eyelid dermatochalasis that overhangs the upper eyelid margin) or
   2. Dermatochalasis that extends less than 3 mm above the upper eyelid margin.
3. Horner syndrome.
4. Marcus Gunn jaw winking syndrome.
5. Myasthenia gravis.
6. Mechanical ptosis, including ptosis due to orbital or lid tumor, cicatricial processes affecting the movements of the upper lid, and enophthalmos.
7. Previous ptosis surgery (previous blepharoplasty [only] is allowed provided the surgery took place > 3 months prior to Visit 1).
8. Lid position affected by lid or conjunctival scarring.
9. Visual field loss from any cause other than ptosis.
10. History of herpes keratitis.
11. History of closed/narrow angle glaucoma (unless patent peripheral iridotomy has been performed > 3 months prior to Visit 1).
12. Periocular neurotoxin (eg, Botox, Xeomin, Dysport, Myobloc) injections within 3 months prior to Visit 1 and during the study.
13. Topical application of bimatoprost (ie, Latisse®) to the eyelashes within 7 days prior to Visit 1 and during the study.
14. Use of topical ophthalmic medications (including anti-allergy [eg, antihistamines], dry eye [ie, Restasis®] and anti-inflammatory drugs [including nonsteroidal anti-inflammatory drugs (NSAIDs) and steroids] other than the assigned study medication within 7 days prior to Visit 1 and during the study. Topical ophthalmic prostaglandin analogues for the treatment of elevated intraocular pressure are permitted if dosed in the evening in accordance with the approved prescribing information. All other topical antiglaucoma medications are prohibited
15. Intravitreal injections (eg, Lucentis®, Eylea®, Avastin®, Triesence®) within 7 days prior to Visit 1 and during the study.
16. Current punctal plugs or placement of punctal plugs during the study.
17. Use of over the counter (OTC) vasoconstrictor/decongestant eye medication (eg, Visine® L.R.®) or any ophthalmic or non-ophthalmic α adrenergic agonist including OTC products (eg, Afrin®) at any time during the study; nonpreserved artificial tears are allowed.

    General
18. Resting heart rate (HR) outside the normal range (60-100 beats per minute).
19. Hypertension with resting diastolic blood pressure (BP) > 105 mm Hg.
20. Use of monoamine oxidase inhibitors (MAOIs; eg, isocarboxazid, phenelzine, tranylcypromine) within 14 days prior to Visit 1 and during the study.
21. Advanced arteriosclerotic disease or history of cerebrovascular accident (CVA).
22. History of hyperthyroidism or thyroid eye disease (ie, exophthalmos, upper eyelid retraction, diplopia secondary to extraocular muscle involvement). Hypothyroidism that is controlled on medication is allowed.
23. Patients with diabetic retinopathy may not be enrolled. However, patients with insulin dependent diabetes, diabetes requiring oral hypoglycemic drugs, or diet controlled diabetes are allowed.
24. Pregnancy or lactation.
25. Diagnosed benign prostatic hypertrophy requiring medicinal therapy; previous prostatectomy is allowed.
26. History of contact or systemic allergic reaction to oxymetazoline or other sympathomimetic drugs (eg, phenylephrine, pseudoephedrine, ephedrine, phenylpropanolamine, fepradinol, or methoxamine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chuck Slonim, MD, Principal Investigator — Oculos Clinical Research
Locations (14):
- United States (14):
  - Artesia, California
  - Newport Beach, California
  - Rancho Cordova, California
  - Santa Maria, California
  - Fort Myers, Florida
  - Largo, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Roswell, Georgia
  - Pittsburg, Kansas
  - Shawnee Mission, Kansas
  - Mason, Ohio
  - Kingston, Pennsylvania
  - Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Planned sample size approx 150 subjects, 100 subjects in the RVL-1201 group, and 50 in the Vehicle group, to be enrolled at approx 20 clinical sites in the US.
Groups:
- RVL-1201: RVL-1201 (oxymetazoline hydrochloride) Ophthalmic Solution 0.1%, one drop each eye QD in the morning
- Vehicle: Vehicle Placebo Ophthalmic Solution, one drop each eye QD in the morning
Period: Overall Study
Arm/Group | RVL-1201 | Vehicle
Started | 94 | 46
Subjects Randomized | 94 | 46
Subjects Treated | 94 | 46
Completed | 90 | 45
Not Completed | 4 | 1
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | RVL-1201 | Vehicle | Total
Number analyzed (Participants) | 94 | 46 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 22 | 60
  >=65 years | 56 | 24 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (12.22) | 63.2 (12.45) | 64.2 (12.28)
Age, Customized [Number; unit: years]
  Median | 68.0 | 65.5 | 67.0
  Minimum | 22 | 26 | 22
  Maximum | 83 | 85 | 85
Sex: Female, Male [Count of Participants; unit: Participants] — Intent to Treat (ITT) Population
  Participants
    Female | 74 | 32 | 106
    Male | 20 | 14 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 11 | 31
  Not Hispanic or Latino | 74 | 35 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 0 | 12
  White | 78 | 3 | 81
  More than one race | 0 | 42 | 42
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 94 | 46 | 140
Iris Color OD (right eye) and Iris Color OS (left eye) [Count of Participants; unit: Participants]
  OD/OS Blue | 23 | 14 | 37
  OD/OS Brown | 55 | 22 | 77
  OD/OS Green | 4 | 1 | 5
  OD/OS Hazel | 12 | 9 | 21
  OD/OS Grey | 0 | 0 | 0
  OD/OS Other | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Number of Points Seen on the Leicester Peripheral Field Test (LPFT) in RVL-1201 Group vs. Vehicle Group
Description: LPFT Total Score is the number of points seen in the top 4 rows on the LPFT. Possible scores range from 0 (no points seen) to 35 (all points seen).
Time Frame: Mean change from Baseline (Day 1, Hour 0) compared with Day 1, Hour 6 and Day 14, Hour 2
Population: Intent-to-Treat (ITT) population: randomized who received at least one dose (total of 140 subjects). Per-Protocol Population (PPP): ITT population with no major protocol deviations (total of 139 subjects). ITT analysis was conducted for the primary endpoint, with Last Observation Carried Forward (LOCF) for missing data.
Measure: Mean (Standard Deviation); unit: Points seen
Groups:
- Vehicle Ophthalmic Solution: Vehicle Placebo Ophthalmic Solution, one drop each eye QD in the morning
Arm/Group | RVL-1201 | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 94 | 46
Points seen
  Mean LPFT-Day 1 Hour 6 | 5.2 (5.97) | 1.5 (3.93)
  Mean LPFT-Day 14 Hour 2 | 6.4 (5.04) | 2.2 (5.80)
Statistical Analysis 1: Comparison: RVL-1201 vs Vehicle Ophthalmic Solution; Test type: Superiority; p < 0.0001, ANCOVA; Two-sided t-test with treatment as a fixed factor and baseline score as a covariate

2. Secondary Outcome: Mean Change From Baseline in Marginal Reflex Distance (MRD) in the Study Eye
Description: MRD is the distance from the center pupillary light reflex to the central margin of the upper eyelid. The MRD is measured from an external photograph.
Time Frame: Baseline Day 1 (Hour 0) and Day 1, Day 14, and Day 42
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters (mm)
Arm/Group | RVL-1201 | Vehicle Ophthalmic Solution
Number analyzed (Participants) | 94 | 46
Millimeters (mm)
  Primary Efficacy - Day 1, Hour 6 | 0.94 (0.924) | 0.67 (1.001)
  Primary Efficacy - Day 14, Hour 2 | 1.09 (0.799) | 0.58 (0.975)
  Post Dose - Day 1, Hour 2 | 0.99 (0.776) | 0.50 (0.803)
  Post Dose - Day 1, Hour 8 | 0.93 (0.958) | 0.70 (0.771)
  Post Dose - Day 14, Hour 6 | 1.03 (0.856) | 0.70 (0.985)
  Post Dose - Day 14, Hour 8 | 0.88 (0.857) | 0.68 (1.023)
  Post Dose - Day 42 | 1.25 (1.036) | 0.79 (1.020)
Statistical Analysis 1: Comparison: RVL-1201 vs Vehicle Ophthalmic Solution; Test type: Superiority; p = 0.12, ANCOVA; Two-sided t-test

ADVERSE EVENTS:
Time Frame: Duration of treatment is 6 weeks (42 Days)
Description: Adverse Events (AEs) spontaneously reported by the subject and/or in response to open-ended questions from study personnel or revealed by observation and are recorded in the Case Report Form (CRF).
Arm/Group | RVL-1201 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/94 | 0/46
Other Adverse Events (participants affected / at risk) | 20/94 | 15/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVL-1201 (N=94) | Vehicle (N=46)
Hyperparathyroidism (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RVL-1201 (N=94) | Vehicle (N=46)
Atrial fibrilation (Cardiac disorders) | 0 (0) | 1 (1)
Punctate keratitis (Eye disorders) | 7 (11) | 2 (2)
Vision blurred (Eye disorders) | 5 (10) | 0 (0)
Ocular hyperaemia (Eye disorders) | 3 (5) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (2)
Dry eye (Eye disorders) | 0 (0) | 1 (2)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (2)
Eye pruritus (Eye disorders) | 0 (0) | 1 (2)
Foreign body sensation (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 0 (0) | 2 (2)
Instillation site pain (General disorders) | 4 (8) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Vital dye staining cornea present (Investigations) | 2 (4) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days